CLINICAL TRIAL: NCT01739764
Title: An Open-Label, Extension (Rollover) Study of Vemurafenib in Patients With BRAF V600 Mutation-Positive Malignancies Previously Enrolled in an Antecedent Vemurafenib Protocol
Brief Title: An Extension (Rollover) Study of Vemurafenib in Participants With BRAF V600 Mutation-Positive Malignancies Previously Enrolled in an Antecedent Vemurafenib Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28399; 2012-003144-80 (EudraCT Number)
Record Dates: First submitted 2012-11-26; First posted 2012-12-03 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vemurafenib 480mg BID (Experimental): Participants received oral vemurafenib at 480 mg BID, depending on the last dose in the antecedent protocol until progression of disease or as long as the participant is deriving clinical benefit, as judged by the investigator, death, withdrawal of consent, unacceptable toxicity, loss to follow-up, or decision of the sponsor to terminate the study, whichever occurs first.
  Interventions: Drug: Vemurafenib
- Vemurafenib 720mg BID (Experimental): Participants received oral vemurafenib at 720 mg BID, depending on the last dose in the antecedent protocol until progression of disease or as long as the participant is deriving clinical benefit, as judged by the investigator, death, withdrawal of consent, unacceptable toxicity, loss to follow-up, or decision of the sponsor to terminate the study, whichever occurs first.
  Interventions: Drug: Vemurafenib
- Vemurafenib 960mg BID (Experimental): Participants received oral vemurafenib at 960 mg BID, depending on the last dose in the antecedent protocol until progression of disease or as long as the participant is deriving clinical benefit, as judged by the investigator, death, withdrawal of consent, unacceptable toxicity, loss to follow-up, or decision of the sponsor to terminate the study, whichever occurs first.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib was given based on the last dose of the antecedent study (minimum 480 mg orally BID).
  Other Names: Zelboraf

SUMMARY:
This open-label, multicenter, non-randomized study provided continued access to vemurafenib for eligible participants with BRAF V600 mutation-positive malignancy, who were previously enrolled and treated in an antecedent vemurafenib protocol and did not meet the protocol's criteria for disease progression, or were treated beyond progression and were still deriving clinical benefit (as assessed by investigator), and may have therefore potentially benefited from continued treatment with vemurafenib. Participants received treatment with oral vemurafenib at 960 milligrams (mg) twice daily (BID), 720 mg BID, or 480 mg BID, depending on the last dose in the antecedent protocol. Treatment continued until progression of disease or as long as the participant was deriving clinical benefit, as judged by the investigator (case-by-case decision with approval of the Medical Monitor), death, withdrawal of consent, unacceptable toxicity, loss to follow-up, or decision of the Sponsor to terminate the study, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* BRAF V600 mutation-positive malignancy
* Prior eligibility for and on study treatment from an antecedent vemurafenib protocol
* Ability to begin treatment in the extension (rollover) protocol within 15 days following the last day of the study in the antecedent protocol
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use 2 adequate methods of contraception as defined by protocol during the course of this study and for at least 6 months after completion of study treatment

Exclusion Criteria:

* Adverse event requiring discontinuation of vemurafenib in the antecedent protocol
* Progressive disease during the antecedent protocol. If approval to treat beyond progression was already given in the antecedent protocol, the participant may roll over into the current protocol without sponsor approval. Under special circumstances, enrollment into this protocol and dosing beyond progression may be considered and will require approval of the sponsor

Participants meeting any of the following exclusion criterion of the antecedent study at the time the participant is considered for the extension (rollover) study:

* Current, recent (within 28 days prior to Day 1), or planned use of any antitumor therapy outside this study
* Any other serious concomitant medical condition that, in the opinion of the investigator, would compromise the safety of the participant or compromise the participant's ability to participate in the study
* History of malabsorption or other clinically significant metabolic dysfunction
* History of clinically significant cardiac or pulmonary dysfunction as specified in antecedent study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-02-19 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (83):
- United States (12):
  - Highlands Oncology Group, Rogers, Arkansas
  - UCLA Department of Medicine, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Chicago Medical Center; Medicine, Section of Pulmonary, Chicago, Illinois
  - Siouxland Regional Cancer Center d/b/a June E. Nylen Cancer Center, Sioux City, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - New York University Medical Center PRIME, New York, New York
  - Evelyn H. Lauder Center, New York, New York
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Mary Crowley Medical Research Center; Oncology, Dallas, Texas
  - M D Anderson Physician Network, Webster, Texas
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- N.N. Alexandrov National Cancer Centre of Belarus, Minsk District, Belarus
- Institut Jules Bordet, Brussels, Belgium
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - University Clinic Centre Sarajevo, Sarajevo
- Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil
- McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec, Canada
- Croatia (2):
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Bank of Cyprus Oncology Center, Nicosia, Cyprus
- Egypt (4):
  - Medical Research Institute, Alexandria
  - National Cancer Institute, Cairo
  - Mansoura University Hospital, Dakahlia
  - Gharbia Cancer Society, Tanta
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz; Apotheke, Mainz
  - Universitätsklinikum Wurzburg, Würzburg
- University General Hospital of Heraklion, Crete, Greece
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Debreceni Egyetem Klinikai Központ; Bőrgyógyászati Klinika, Debrecen
  - Pecsi Tudomanyegyetem, Pécs
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center; Allergy and Clinical Immunology Unit, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Maastricht University Medical Center, Maastricht, Netherlands
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Clinical Studies Trust, Christchurch
- Portugal (2):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Medisprof SRL, Cluj-Napoca, Romania
- Russia (6):
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin"; Chemotherapy Departement, Moskva, Moscow Oblast
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan'
  - SBIH " Clinical Oncological Dispensary # 1"; Chemotherapy department #1 and #2, Krasnodar
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - St. Petersburg SHI "City Clinical Oncology Dispensary", Saint Petersburg
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
- South Africa (3):
  - Cape Town Oncology Trials, Cape Town
  - Wits Donald Gordon Clinical Trial Centre; Medical Oncology, Parktown, Johannesburg
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth
- South Korea (5):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (16):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Regional Universitario de Malaga; Oncologia, Málaga, Malaga
  - Hospital General Universitario Santa Lucia, Cartagena (Murcia), Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (3):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Churchill Hospital, Oxford
  - Royal Marsden Hospital, Surrey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 82 centers in 24 countries.
Pre-assignment Details: 215 participants were enrolled into this OLE study and were included in the Safety population.
Period: Overall Study
Arm/Group | Vemurafenib 480mg BID | Vemurafenib 720mg BID | Vemurafenib 960mg BID
Started | 29 | 40 | 146
Completed | 3 | 4 | 20
Not Completed | 26 | 36 | 126
Not completed — Adverse Event | 0 | 3 | 4
Not completed — Death | 4 | 6 | 38
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Non-Compliance | 0 | 0 | 1
Not completed — Multiple Reasons | 3 | 2 | 3
Not completed — Physician Decision | 2 | 2 | 4
Not completed — Progressive Disease | 3 | 5 | 16
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Study Terminated by Sponsor | 8 | 13 | 26
Not completed — Withdrawal by Subject | 6 | 5 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib 480mg BID | Vemurafenib 720mg BID | Vemurafenib 960mg BID | Total
Number analyzed (Participants) | 29 | 40 | 146 | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (11.7) | 60.6 (12.4) | 52.3 (13.5) | 54.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 57 | 95
  Male | 11 | 20 | 89 | 120
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 2 | 2 | 3 | 7
    Not Hispanic or Latino | 24 | 37 | 137 | 198
    Not Stated | 0 | 0 | 1 | 1
    Unknown | 3 | 1 | 5 | 9
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Asian | 2 | 2 | 39 | 43
    Black or African American | 1 | 0 | 0 | 1
    White | 23 | 37 | 101 | 161
    Other | 0 | 1 | 2 | 3
    Unknown | 3 | 0 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Intensity of Vemurafenib
Description: Dose Intensity was defined as (total actual doses taken/total planned doses) *100, where total planned doses = prescribed doses * planned days on treatment, where planned days on treatment were defined as the interval between date of first dose and date of last dose.
Time Frame: Baseline up to a maximum of 7 years.
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study medication. Please note that for this Outcome Measure, one participant who received 960 mg BID of Vemurafenib had no treatment end date indicated and was excluded from the calculation of study treatment exposure summaries.
Measure: Mean (Standard Deviation); unit: Percentage of Planned Dose
Arm/Group | Vemurafenib 480mg BID | Vemurafenib 720mg BID | Vemurafenib 960mg BID
Number analyzed (Participants) | 29 | 40 | 145
Percentage of Planned Dose | 95.3 (8.1) | 92.9 (12.1) | 94.5 (11.0)

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events. Reported are the Percentage of Participants with AEs and Serious Adverse Events (SAEs).
Time Frame: Baseline up to 28 days after the last dose of study drug (up to a maximum of 7 years).
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vemurafenib 480mg BID | Vemurafenib 720mg BID | Vemurafenib 960mg BID
Number analyzed (Participants) | 29 | 40 | 146
Percentage of Participants
  AEs | 93.1 | 92.5 | 93.2
  SAEs | 48.3 | 37.5 | 19.9

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose of study drug (up to a maximum of 7 years).
Arm/Group | Vemurafenib 480mg BID | Vemurafenib 720mg BID | Vemurafenib 960mg BID
All-Cause Mortality (participants affected / at risk) | 4/29 | 6/40 | 38/146
Serious Adverse Events (participants affected / at risk) | 14/29 | 15/40 | 29/146
Other Adverse Events (participants affected / at risk) | 21/29 | 29/40 | 119/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib 480mg BID (N=29) | Vemurafenib 720mg BID (N=40) | Vemurafenib 960mg BID (N=146)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
CATARACT NUCLEAR (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
PAROPHTHALMIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TRACHEAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MYOPATHY TOXIC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BRAIN NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (4)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
TRACHEAL RESECTION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib 480mg BID (N=29) | Vemurafenib 720mg BID (N=40) | Vemurafenib 960mg BID (N=146)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 5 (6) | 13 (18)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
UVEITIS (Eye disorders) | 2 (2) | 2 (5) | 3 (4)
VISION BLURRED (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (6) | 4 (4) | 4 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 3 (6) | 3 (5) | 16 (18)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 8 (8)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 8 (8) | 16 (22)
VOMITING (Gastrointestinal disorders) | 2 (2) | 4 (5) | 12 (13)
ASTHENIA (General disorders) | 3 (4) | 5 (5) | 3 (3)
FATIGUE (General disorders) | 2 (2) | 5 (5) | 28 (33)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2) | 5 (6)
PYREXIA (General disorders) | 1 (1) | 1 (2) | 9 (11)
CHORIORETINITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1) | 10 (10)
PNEUMONIA (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 1 (1) | 6 (7)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 4 (5) | 1 (1)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 6 (8)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (3) | 3 (4)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 4 (9) | 8 (8)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 2 (2) | 1 (2)
BLOOD CREATININE INCREASED (Investigations) | 1 (3) | 3 (3) | 8 (10)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 2 (2) | 7 (11)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1) | 10 (10)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 19 (24)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (15) | 30 (41)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 9 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 6 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 7 (12)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4) | 3 (3)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (2) | 4 (5)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 16 (24)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 7 (13)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 4 (4) | 15 (15)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 10 (10)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 7 (12)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 21 (21)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 9 (10)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 7 (13)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 20 (21)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 12 (13)
PANNICULITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (10)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 22 (32)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 13 (15)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 14 (16)
HYPERTENSION (Vascular disorders) | 2 (2) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT01739764/Prot_SAP_000.pdf